CLINICAL TRIAL: NCT04843878
Title: Feasibility Testing of a New COVID-19 Testing Platform
Brief Title: COVID-19 Testing Pilot Study
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Benjamin S. Abella, MD, MPhil (Unknown); Marcelo Der Torossian Torres, Ph.D. (Unknown); Cesar De La Fuente, Ph.D. (Unknown)
Responsible Party: Sponsor
Other Study IDs: 844488
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Diagnostic Test, Routine; Coronavirus; Diagnoses Disease; Rapid Coronavirus Test
Keywords: COVID-19; Detect; Pandemic; Symptomatic; Asymptomatic; Anterior Nares
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive: Subjects that tested positive for COVID-19 based on the clinical gold standard PCR test.
  Interventions: Diagnostic Test: COVID Detect
- Negative: Subjects that tested negative for COVID-19 based on the clinical gold standard PCR test.
  Interventions: Diagnostic Test: COVID Detect

INTERVENTIONS:
Diagnostic Test: COVID Detect — The study is determining the efficacy of a new rapid COVID testing method.

SUMMARY:
The purpose of this study is to determine the reliability of a low-cost rapid diagnostic test for COVID-19. The method of the testing procedure uses electrochemistry to detect COVID-19 spike proteins within human samples. To test the effectiveness of this new method, patients will be recruited as they present for testing at ambulatory Penn testing sites. Patients will be asked to self-collect one anterior nares samples under the supervision of authorized study personnel.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be an adult (age>17) and either sex.
2. Written informed consent must be obtained prior to study enrollment.

   a. A subject who is eighteen (18) years or older must be willing to give written informed consent and must agree to comply with study procedures.
3. Subject must be able to read and write in English.

Exclusion Criteria:

1. The subject is currently receiving or has received within the past thirty (30) days of the study visit an experimental biologic, drug, or device including either treatment or therapy.
2. The subject has previously participated in this research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited as they present for treatment at ambulatory Penn testing sites. Subjects who present with symptoms of COVID-19-like illness at the study site as defined in Inclusion Criteria below and have come to the study site for routine evaluation of their condition may be enrolled in this clinical study. Males and females aged >17 years old may be enrolled, and should be represented in proportions representative of the population.
Sampling Method: Non-Probability Sample
Enrollment: 326 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-12 (Actual)

PRIMARY OUTCOMES:
Device Accuracy - Positive and Negative Percentage | 3 Months
  The accuracy of the new prototype testing method will be determined by comparing the prototype's result to the clinical gold standard PCR test. The accuracy will be determined by calculating the percentage of the test's ability to correctly identify both the presence and absence of virus compared to the PCR result for the positive and negative results.
Device Accuracy - False positive and False negative percentage | 3 Months
  The accuracy of the test will also be determined based on the percentage of false-positives and false-negatives compared to the gold standard clinical PCR test.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin S Abella, MD, MPhil, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD.